CLINICAL TRIAL: NCT01687023
Title: A Wearable System to Monitor Tai Chi Practice
Status: Completed | Type: Observational
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Other Study IDs: 2011-P-001597
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Tai Chi; Wearable sensors; Movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tai Chi: Healthy Tai Chi practitioners

SUMMARY:
The goal of this research study is to show that features derived from data gathered using SHIMMER wearable sensor platform can capture adherence and proficiency in the performance of exercises that are part of Tai Chi interventions.

ELIGIBILITY:
Inclusion Criteria:

* Young style Tai Chi practitioners

Exclusion Criteria:

* Any movement impairment that will impede Tai Chi movements performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Tai Chi practitioners in a wide range of proficiency
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Biomarkers of adherence and proficiency | 1 day
  Data gathered using SHIMMER devices will be segmented to derive signal features. These features will be then used to feed a pattern recognition algorithm the output of which indicates whether a specific Tai Chi movement of interest has been performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States